CLINICAL TRIAL: NCT05686421
Title: A Single-Center Proof Of Concept Study of a Novel Comfortable and Stabilizing Chin & Forehead Rest Attachment for Slit Lamp Configuration Devices
Brief Title: Comfortable and Stabilizing Chin & Forehead Rest Attachment for Slit Lamp Configurations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped prior to collection of data from participants due to investigator transfer.
Sponsor: NYU Langone Health (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-01420
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Age-Related Macular Degeneration; Diabetic Retinopathy; Central Serous Chorioretinopathy; Glaucoma; Glaucoma, Suspect; Eye Diseases
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Central Serous Chorioretinopathy; Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Device C (OD-OS), then Device N (OD-OS) (Experimental): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device C, a standard conventional device with no attachment; and device N, the standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device.
  Participants will first be imaged using device C starting with the right eye (OD), then left eye (OS). They will then be imaged using device N, starting with OD, then OS.
  Interventions: Device: OCT Imaging Using Device N; Device: OCT Imaging Using Device C
- Device C (OS-OD), then Device N (OS-OD) (Experimental): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device C, a standard conventional device with no attachment; and device N, the standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device.
  Participants will first be imaged using device C starting with the left eye (OS), then right eye (OD). They will then be imaged using device N, starting with OS, then OD.
  Interventions: Device: OCT Imaging Using Device N; Device: OCT Imaging Using Device C
- Device N (OD-OS), then Device C (OD-OS) (Experimental): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device N, a standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device; and device C, the standard conventional device with no attachment.
  Participants will first be imaged using device N starting with the right eye (OD), then left eye (OS). They will then be imaged using device C, starting with OD, then OS.
  Interventions: Device: OCT Imaging Using Device N; Device: OCT Imaging Using Device C
- Device N (OS-OD), then Device C (OS-OD) (Experimental): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device N, a standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device; and device C, the standard conventional device with no attachment.
  Participants will first be imaged using device N starting with the left eye (OS), then right eye (OD). They will then be imaged using device C, starting with OS, then OD.
  Interventions: Device: OCT Imaging Using Device N; Device: OCT Imaging Using Device C

INTERVENTIONS:
Device: OCT Imaging Using Device N — Standard conventional OCT imaging device equipped with extendable and comfortable chin and forehead rest.
Device: OCT Imaging Using Device C — Standard conventional OCT imaging device.

SUMMARY:
In this study, participants will be imaged using two Optical Coherence Tomography (OCT) devices: device N, a standard conventional OCT device with an invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device; and device C, the standard conventional OCT device with no invention attached. The investigators will assess whether the chin and forehead rest attachment (invention) provides a more comfortable experience for patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers; OR,
* AMD, diabetic retinopathy, central serous chorioretinopathy, and/or glaucoma or glaucoma suspects or any other suspected eye disease

Group-Specific Inclusion Criteria:

-- There are no group-specific inclusion criteria for patients with AMD, diabetic retinopathy, and central serous chorioretinopathy.

Healthy Volunteers

* A normal clinical ophthalmic examination.
* Reliable VF, reproducible glaucoma hemifield tests labeled within normal limits on at least one test.
* Good quality (adequate signal strength ≥ 6/10, without segmentation algorithm failure and motion artifacts > 1 vessel diameter) RNFL and Ganglion Cell Inner Plexiform Layer (GCIPL) OCT, within normal limits.

Primary Open Angle Glaucoma (POAG)

* Clinical characteristics of glaucoma: optic nerve head (ONH) abnormalities: global rim thinning, rim notch, or disc hemorrhage; retinal nerve fiber layer (RNFL) defect.
* Typical glaucomatous field loss in reliable VF, reproducible glaucoma hemifield tests labeled outside normal limits on at least two consecutive tests.
* Good quality (adequate signal strength ≥ 6/10, without segmentation algorithm failure and motion artifacts > 1 vessel diameter) RNFL and GCIPL OCT, labeled outside normal limits with typical glaucomatous RNFL and GCIL thinning.

Normal Tension Glaucoma (NTG)

* Identical to POAG criteria with IOP recorded at ≤ 21 mmHg at any time point.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

- Any medical treatment (e.g., chronic corticosteroid, hydroxychloroquine, chloroquine, thioridazine, canthaxanthine) or conditions that affect VF (e.g., stroke) and retinal thickness other than glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Gadi Wollstein, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Gadi.Wollstein@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access to the data upon reasonable request. Requests should be directed to Gadi.Wollstein@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Device C (OD-OS), Then Device N (OD-OS): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device C, a standard conventional device with no attachment; and device N, the standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device.
  Participants will first be imaged using device C starting with the right eye (OD), then left eye (OS). They will then be imaged using device N, starting with OD, then OS.
  OCT Imaging Using Device N: Standard conventional OCT imaging device equipped with extendable and comfortable chin and forehead rest.
  OCT Imaging Using Device C: Standard conventional OCT imaging device.
- Device C (OS-OD), Then Device N (OS-OD): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device C, a standard conventional device with no attachment; and device N, the standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device.
  Participants will first be imaged using device C starting with the left eye (OS), then right eye (OD). They will then be imaged using device N, starting with OS, then OD.
  OCT Imaging Using Device N: Standard conventional OCT imaging device equipped with extendable and comfortable chin and forehead rest.
  OCT Imaging Using Device C: Standard conventional OCT imaging device.
- Device N (OD-OS), Then Device C (OD-OS): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device N, a standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device; and device C, the standard conventional device with no attachment.
  Participants will first be imaged using device N starting with the right eye (OD), then left eye (OS). They will then be imaged using device C, starting with OD, then OS.
  OCT Imaging Using Device N: Standard conventional OCT imaging device equipped with extendable and comfortable chin and forehead rest.
  OCT Imaging Using Device C: Standard conventional OCT imaging device.
- Device N (OS-OD), Then Device C (OS-OD): Participants will be randomized to receive 1 macular scan on each eye and 1 optic nerve head (ONH) scan on each eye from two devices: device N, a standard conventional device with the invention (comfortable chin and forehead rest that can be adjusted to fit each individual's size) attached to the device; and device C, the standard conventional device with no attachment.
  Participants will first be imaged using device N starting with the left eye (OS), then right eye (OD). They will then be imaged using device C, starting with OS, then OD.
  OCT Imaging Using Device N: Standard conventional OCT imaging device equipped with extendable and comfortable chin and forehead rest.
  OCT Imaging Using Device C: Standard conventional OCT imaging device.
Period: Overall Study
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Started | 42 | 0 | 0 | 0
Completed | 20 | 0 | 0 | 0
Not Completed | 22 | 0 | 0 | 0
Not completed — Screen failure | 22 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the "Device C (OS-OD), then Device N (OS-OD)", "Device N (OD-OS), then Device C (OD-OS)", or "Device N (OS-OD), then Device C (OS-OD)" arm due to termination of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD) | Total
Number analyzed (Participants) | 42 | 0 | 0 | 0 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.42 (18.83) |  |  |  | 60.42 (18.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 |  |  |  | 30
  Male | 12 |  |  |  | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 |  |  |  | 9
  Not Hispanic or Latino | 25 |  |  |  | 25
  Unknown or Not Reported | 8 |  |  |  | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 5 |  |  |  | 5
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 4 |  |  |  | 4
  White | 23 |  |  |  | 23
  More than one race | 2 |  |  |  | 2
  Unknown or Not Reported | 8 |  |  |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 42 |  |  |  | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Indicate Device N Provided a More Comfortable Experience, Compared With Device C
Description: Participants will be asked which device provided a more comfortable experience: Device C or Device N.
Time Frame: Post-Imaging Session (Day 1)
Population: N=0 participants were analyzed in the "Device C (OD-OS), then Device N (OD-OS)" arm due to early termination of the trial prior to data collection from participants. N=0 participants were analyzed in the "Device C (OS-OD), then Device N (OS-OD)", "Device N (OD-OS), then Device C (OD-OS)," and "Device N (OS-OD), then Device C (OS-OD)" arms because no participants were enrolled into these arms.
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Comfort Level Rating of Device N on 0-5 Scale
Description: Participants will be asked to rate how comfortable Device N was, on a scale of 0-5. Higher scores indicate higher levels of comfort.
Time Frame: Post-Imaging Session (Day 1)
Population: as for outcome 1
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Comfort Level Rating of Device C on 0-5 Scale
Description: Participants will be asked to rate how comfortable Device C was, on a scale of 0-5. Higher scores indicate higher levels of comfort.
Time Frame: Post-Imaging Session (Day 1)
Population: as for outcome 1
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Time Duration to Adjust for Number of Motion Artifacts Present With Device N Imaging
Description: The OCT imaging device includes an "eye tracking" feature that selects a specific location within the eye and constantly adjusts, i.e. tracks, for fine fixation adjustments that occur when a patient's eye is moving very slightly during imaging. The time to adjust for the number of motion artifacts present will be defined as the duration it takes from the moment the imager clicks "Acquire" on the device to when the progress bar is "Full."
Time Frame: Imaging Session (Day 1)
Population: as for outcome 1
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time Duration to Adjust for Number of Motion Artifacts Present With Device C Imaging
Description: as for outcome 4
Time Frame: Imaging Session (Day 1)
Population: as for outcome 1
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: N/A - no participants were assessed for adverse events.
Description: N/A - no participants were assessed for adverse events.
Arm/Group | Device C (OD-OS), Then Device N (OD-OS) | Device C (OS-OD), Then Device N (OS-OD) | Device N (OD-OS), Then Device C (OD-OS) | Device N (OS-OD), Then Device C (OS-OD)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT05686421/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT05686421/ICF_000.pdf